CLINICAL TRIAL: NCT02569216
Title: Electrical Inhibition (EI): A Preliminary Study To Prevent The Uterine Contractions Of Human Preterm Labor And Preterm Birth
Brief Title: Electrical Inhibition (EI): A Preliminary Study To Inhibit Preterm Labor And Preterm Birth
Acronym: EI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA/IRB approved but hospital administration vetoed the study fearing litigation of a preterm birth though the electrical uterine pacemaker/EI is not the cause.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-00553; G080036 (Other: FDA)
Record Dates: First submitted 2015-10-01; First posted 2015-10-06 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Premature Birth; Premature Labor
Keywords: Electrical Inhibition; Preterm Birth; Premature Birth; Preterm Labor; Premature Labor; tocolytic; uterus
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Electrical Inhibition (EI) intervention (Experimental): Electrical Inhibition (EI) uterine pacemaker is activated only when there is a preterm uterine contraction. The EI uterine pacemaker delivers a 1-15mA (20mA maximum) constant direct current for only 2 seconds only while there is a preterm uterine contraction.
  Interventions: Device: Electrical Inhibition (EI)

INTERVENTIONS:
Device: Electrical Inhibition (EI) — constant direct current 1-20mA transvaginal 10 second bursts only when needed

SUMMARY:
An electrical-inhibition (EI) uterine pacemaker device similar to an electrical heart pacemaker delivers a weak electrical current to the human uterus during active preterm labor to rapidly and safely inhibit the unwanted premature uterine contractions and possibly a preterm birth.

DETAILED DESCRIPTION:
Electrical intervention (EI) uses bipolar, constant-current (1-20 mA), square-wave pulses in 20% duty cycles. Women in active preterm labor have an electrode catheter placed into the posterior fornix of the vaginal canal. The EI current is given up to 80 minutes while monitoring tocodynamometric (toco) contractions and adjunct electrohysterographic (EHG) activity while continuously monitoring maternal vital signs, fetal heart rate and electrocardiogram (fECG). The study includes a pre-EI control period (C1); the EI period, when a 10-second current burst is delivered only during a contraction; and a post-EI control period (C2). The whole study will take a maximum of two hours.

The uterine toco contraction frequency and adjunct EHG electrical activity are analyzed for changes caused by EI. Changes in maternal vital signs, fetal heart rate and fECG will determine EI side-effects.

ELIGIBILITY:
Inclusion Criteria:

* between 24 to 34 weeks pregnant with a singleton gestation;
* in preterm labor as defined by the American College of Obstetricians and Gynecologists and the American Academy of Pediatrics,78 as follows:

  * persistent uterine contractions (4 every 20 minutes or 8 every 60 minutes)
  * And any one or more of the following:

    * Documented cervical change
    * > 1cm cervical dilatation and progressing
    * > 80% cervical effacement
* anticipate a normal spontaneous vaginal delivery (NSVD).
* at least 18 years of age
* signed a written Informed Consent Document
* willing and able to comply with study requirements

Exclusion Criteria:

* severe preeclampsia
* severe abruption placenta
* rupture of amniotic membranes
* frank chorioamnionitis
* fetal death
* fetal anomaly incompatible with life
* severe fetal growth restriction (EFW <5%)
* mature fetal lung studies
* maternal cardiac arrhythmias
* a permanent cardiac pacemaker
* a fetal cardiac arrhythmia
* contraindication for tocolysis

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Decrease tocodynamometric monitored preterm uterine contraction frequency | 30 seconds
  Measure changes in preterm uterine mechanical contraction frequency as assessed by the tocodynamometer. This will be done for the duration of the study.

SECONDARY OUTCOMES:
Decrease adjunct electrohysterographic monitored preterm uterine contraction electrical activity. | 20 seconds
  Measure changes in preterm uterine electrical contraction activity as assessed by the electrohysterogram. This will be done for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Karsdon, M.D., Study Director — New York University Hospital
Locations (1):
- New York University Hospital, Manhattan, New York, United States

REFERENCES:
- [Result] Karsdon J, Garfield RE, Shi SQ, Maner W, Saade G. Electrical inhibition of preterm birth: inhibition of uterine contractility in the rabbit and pup births in the rat. Am J Obstet Gynecol. 2005 Dec;193(6):1986-93. doi: 10.1016/j.ajog.2005.05.009. PMID 16325601
- [Result] Karsdon J, El Daouk M, Huang WM, Ashmead GG. Electrical pacemaker as a safe and feasible method for decreasing the uterine contractions of human preterm labor. J Perinat Med. 2012 Nov;40(6):697-700. doi: 10.1515/jpm-2012-0136. PMID 23089601